CLINICAL TRIAL: NCT05279352
Title: A Two-stage Randomized, Placebo-controlled, Double-blind, Phase 2a Study to Characterize the Safety and Pharmacokinetics of FBR-002 in Patients Hospitalized With COVID-19 in Need of Supplemental Oxygen and at Risk of Severe Outcome
Brief Title: Safety and Pharmacokinetics of FBR-002 for the Treatment of Patients Hospitalized With COVID-19 in Need of Supplemental Oxygen and at Risk of Severe Outcome
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fab'entech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: E21-04
Record Dates: First submitted 2022-03-14; First posted 2022-03-15 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — FBR-002

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Arm (Experimental): FBR-002 at 4.3 EU/kg on D1 and D3 or FBR-002 at 5.7 EU/kg on D1 and D3
  Interventions: Drug: FBR-002
- Placebo Arm (Placebo Comparator): Two administrations of placebo at D1 and D3
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: FBR-002 — Administration on D1 and D3
  Arms: Treatment Arm
Drug: Placebo — Administration on D1 and D3
  Arms: Placebo Arm

SUMMARY:
Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) is the coronavirus associated with COVID-19 (Coronavirus Disease 2019), invading the respiratory tract, and leading to symptoms from dysgeusia, anosmia, fever, headache and cough to dyspnea and severe respiratory failure and even death. In order to obtain its pathogenic activity, the SARS-CoV-2 relies on its spike protein to enter the cells of the infected patient. This infection leads to a variable severity spectrum, with the majority of forms of mild entity (upper respiratory tract infection or lower respiratory tract without respiratory failure or insufficiency of other organs) despite the presence of a considerable share of severe infections in need hospitalization in sub-intensive or intensive area (up to 6% of cases) with invasive and non-invasive respiratory support. Approximately 14% of patients have experienced severe disease and 5% have been critically ill.

In the context of global pandemic, Fab'entech is currently developing polyclonal F(ab')2 equine fragments directed against the SARS-CoV-2 spike protein. Indeed, as virus entry within the cell requires this protein, Fab'entech proposes a way to block this event, neutralizing viral replication, and therefore inhibiting pathogenic activity of the virus.

The objective of this two-stage randomized, placebo-controlled, double blind, phase 2a study is to characterize the safety and pharmacokinetics of FBR-002 in patients hospitalized with COVID-19 in need of supplemental oxygen and at risk of severe outcome

ELIGIBILITY:
Inclusion Criteria:

* I1. Male or female ≥ 18 years
* greater than or equal to 70 years of age with or without any risk factor
* or less than 70 years of age and the presence of at least one of the following risk factors:

  * Arterial hypertension under treatment (all stages)
  * Obesity (body mass index [BMI] ≥30 kg/m²) or severe obesity (BMI of ≥40 kg/m²)
  * Diabetes (all types)
  * Heart conditions (such as heart failure, coronary artery disease, cardiomyopathies or hypertension)
  * Stroke or cerebrovascular disease History
  * Chronic lung diseases, including COPD (chronic obstructive pulmonary disease), asthma (moderate-to-severe), interstitial lung disease, cystic fibrosis, and pulmonary hypertension
  * Malignancies (solid tumors or blood malignancies) that are progressive or were diagnosed less than 5 years ago
  * Immunocompromised state (this includes patients who are suffering from primary immunodeficiencies; patients under treatment with corticosteroids either oral or parenteral; patients receiving active chemotherapy; patients on biological treatment or treatment with Janus Kinase (JAK) inhibitors)
  * Solid organ or blood stem cell transplant
  * Down syndrome
  * Known human immunodeficiency virus (HIV) infection
  * Liver disease of stage 1 and 2 based on the Child-Pugh classification (Appendix C)
  * Hemoglobin blood disorders (Thalassemia, Sickle Cell Disease, etc)
  * Renal disease (grade 1 and 2 according to Kidney Disease Improving Global Outcomes (KDIGO) classification) (see Appendix D)
  * Dementia or other neurological conditions
  * Absence of anti-SARS-CoV2 IgM or IgG at screening
* I2. Written informed consent provided by the patient or by a legal representative
* I3. Biologically confirmed SARS-CoV-2 infection ≤ 10 days before screening
* I4. First onset of COVID-19 symptoms ≤ 10 days, among fever and/or chills, headache, myalgias, cough, shortness of breath, fatigue, the new loss of taste or smell
* I5. Findings in chest-X-ray or chest computed tomography compatible with lower respiratory tract infection* * precision for imaging: typical imaging features related to COVID-19
* I6. Patient admitted to hospital for COVID-19, but outside of the Intensive Care Unit
* I7. Patient requiring low-flow O2 supplementation ≤ 6L/min by mask or nasal prongs at screening
* I8. The score of 5 on the WHO 11-point Clinical Progression Scale at screening

Exclusion Criteria:

* E1. Score ≥ 6 on the WHO 11-point Clinical Progression Scale at screening
* E2. Respiration rate > 30 breaths/min in adults under low-flow (⩽ 6 L/min) oxygen
* E3. Liver failure of stage 3 according to the Child-Pugh classification
* E4. Severe renal failure (≥ grade 3 according to KDIGO classification)
* E5. Treatment with anti-SARS-CoV-2 immunoglobulins or any blood-derived products in the last 90 days
* E6. Any anti-SARS-CoV-2 vaccine injection performed less than 21 days before screening
* E7. Pregnancy or lactation. Women of child-bearing potential will be screened by a urine pregnancy test before inclusion in the study
* E8. Known allergy or hypersensitivity or intolerance to study product components
* E9. History of anaphylaxis during a prior administration of equine serum (i.e., anti- tetanus serum or anti-ophidic serum or anti-arachnid toxin serum or anti-rabies serum) or allergic reaction due to contact or exposure to horses
* E10. Participation in any other Interventional study with an investigational product in the last 30 days or within 5 half-lives of receiving the investigational product
* E11. Patients with short life expectancy or with any severe concomitant illness(es) that, in the Investigator's judgment, would adversely affect the patient's participation in the study
* E12. Septic shock

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-03-21 (Actual); Primary Completion 2022-06-15 (Estimated); Study Completion 2022-07-15 (Estimated)

PRIMARY OUTCOMES:
Adverse events of FBR-002 | Day 1 to Day 14
  The rate of treatment-emergent adverse events (serious and non-serious) of FBR-002 in the two groups of treated patients and vs. placebo over 14 days

SECONDARY OUTCOMES:
Pharmacokinetics of FBR-002 | Day 1 to Day 14
  To characterize the pharmacokinetics (PK) profile of FBR-002 on SARS-CoV-2 infected patients over time from Day D1 to D14, including the mean plasmatic concentration of FBR002 of at least 2.6 μg/mL between Day 1 and Day 7 in treated groups;
Biomarkers | Day 1 to Day 14
  The comparison of the relative changes of biomarkers over the time from D1 to D14 between patients treated with placebo and patients treated with each of the two dose regimens of FBR-002
Viral load | From Day 1 to Day 14
  The comparison of viral load over the time from D1 to D14 between patients treated with placebo and patients treated with each of the two dose regimens of FBR-002
Efficacy of FBR-002 | Day 8
  The comparison of the rate of patients progressing into WHO-CPS ≥6 by Day 8 between patients treated with placebo and patients treated with either dose of FBR-002
Efficacy of FBR-002 | Day 8
  The comparison of the rate of patients with an improvement of at least two points based on the WHO 11-point ordinal CPS i.e., hospital discharge between patients treated with placebo and patients treated with either dose of FBR-002; this is censored at 7 days after the administration of the first dose (Day 8).

CONTACTS AND LOCATIONS:
Overall Officials: Evangelos Giamarellos-Bourboulis, Prof, Principal Investigator — University General Hospital of Athens ATTIKON
Locations (6):
- Greece (6):
  - University General Hospital of Alexandroupolis, Alexandroupoli
  - "Sotiria" General Hospital of Chest Diseases of Athens, Athens
  - University General Hospital of Athens ATTIKON, Athens
  - University General Hospital of Patras, Pátrai
  - "Tzaneio" General Hospital of Piraeus, Piraeus
  - AHEPA University General Hospital of Thessaloniki, Thessaloniki

REFERENCES:
- [Background] Herbreteau CH, Jacquot F, Rith S, Vacher L, Nguyen L, Carbonnelle C, Lotteau V, Jolivet M, Raoul H, Buchy P, Saluzzo JF. Specific polyclonal F(ab')2 neutralize a large panel of highly pathogenic avian influenza A viruses (H5N1) and control infection in mice. Immunotherapy. 2014;6(6):699-708. doi: 10.2217/imt.14.40. Epub 2014 Mar 27. PMID 24673720